CLINICAL TRIAL: NCT05444309
Title: Ultrasound Guided Pericapsular Nerve Group Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Pediatric Hip Surgeries
Brief Title: Ultrasound Guided Pericapsular Nerve Group Block Versus Quadratus Lumborum Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Rehab Abd-Allah Wahdan, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-6-2022
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Pediatric Postoperative Pain
Keywords: Pericapsular Nerve Group Block; Quadratus Lumborum Block; postoperative analgesia; pediatric hip surgeries

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into three equal groups
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadratus lumborum block group (Active Comparator): The child will be positioned in the lateral position, with the operative side non-dependent. Under complete aseptic precautions, QL block will be given by anterior approach at the level of L4. A linear high-frequency probe of Sonosite M Turbo ultrasonography will be applied vertically above the iliac crest, and a 22G, 80 mm spinal needle will be inserted in the plane from the posterior edge of the probe through the QL muscle in an anteromedial direction. The needle tip will be placed between the Psoas major (PM) muscle and the QL muscle.
  After negative aspiration, injection of 0.5 mL of normal saline to the space between PM and QL muscles .
  An injection of 0.5 mg/kg of 0.25% bupivacaine into the fascial plane and the local anesthetic appears to press down the PM muscle in the ultrasound image, the patients will be repositioned to a supine position immediately after the block.
  Interventions: Procedure: Quadratus lumborum (QL) block group
- Pericapsular Nerve Group (PENG) block group (Active Comparator): PENG block will be done while the child in supine position. Then, a high-frequency (8-15 MHz) ultrasound linear probe of Sonosite M Turbo ultrasonography (FUJIFILM Sonosite, Inc., Bothell, WA, USA) will be placed over the anterosuperior iliac spine and then rotating it 45 degrees to acquire images from lateral to medial of the anterior inferior iliac spine, iliopubic eminence, psoas tendon, and the femoral artery.
  Then, a 22G, 80 mm spinal needle will be inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly.
  After negative aspiration and a test does (0.5 mL of normal saline), an injection of 0.5 mg/kg of 0.25% bupivacaine into the space between the psoas tendon and the iliopubic eminence.
  Interventions: Procedure: Pericapsular Nerve Group (PENG) block group
- control group (No Intervention): The child will not receive any block.

INTERVENTIONS:
Procedure: Quadratus lumborum (QL) block group — patient will receive 0.5 mg/kg of bupivacaine 0.25% through the quadratus lumborum block approach
  Other Names: Group Q
  Arms: Quadratus lumborum block group
Procedure: Pericapsular Nerve Group (PENG) block group — patient will receive 0.5 mg/kg of bupivacaine 0.25% through the Pericapsular Nerve Group (PENG) block
  Other Names: Group P
  Arms: Pericapsular Nerve Group (PENG) block group

SUMMARY:
Hip surgeries in pediatrics consider as one of the common nowadays surgeries with sever postoperative pain so pain management is essential to decrease postoperative complications, early mobilization and hospital discharge. Traditional use of opioids is associated with many adverse effects such as sedation, dizziness, nausea, vomiting, constipation and respiratory depression.

Previous studies reported that Quadratus Lumborum (QL) Block and Pericapsular Nerve Group (PENG) Block are effective postoperative analgesia in hip surgeries.

In this study we will compare between QL block and PENG Block for effective postoperative analgesia to reduce opioids consumption and subsequently avoid opioid-related adverse effects, early mobilization and early hospital discharge.

DETAILED DESCRIPTION:
Developmental dysplasia of the hip (DDH) is a common disease of the pediatrics patients with a rate of incidence 3 to 5 per 1000 children and open surgical reduction of congenital hip dislocation (CHD) is commonly done in paediatrics.

One of the most important challenges in pediatric hip surgeries is postoperative pain management which may result in impaired patient rehabilitation and prolonged hospitalizations.

Opioids are commonly used for postoperative analgesia in various surgeries but their use is associated with many complications such as sedation, dizziness, nausea, vomiting, constipation and respiratory depression. Many types of peripheral nerve blocks, such as the femoral nerve block (FNB) and the lumbar plexus block (LPB), are used for lower limb surgeries as well as anterior quadratus lumborum block (QLB) and Pericapsular nerve group (PENG) block that provide effective postoperative analgesia in lower limb surgeries.

Quadratus Lumborum (QL) block was first described by Rafael Blanco at the 2007 annual meeting of the European Society of Regional Anesthesia (ESRA). The basic concept of the QL block is the deposition of a local anesthetic solution adjacent to the anterolateral aspect of the QL muscle. The spread pattern obtained is similar to that of the landmark-based TAP block, in that there is subsequent extension into the thoracic paravertebral space. Borglum et al. originally described placing the needle tip anterior to the QL muscle using their transmuscular approach.

This technique was later refined by applying a posterior approach, named the "Shamrock method" (with the erector spinae, QL, and psoas muscles as the leaves and the L4 transverse process as the stem). Administering local anesthesia between the QL and psoas muscles ensures a reliable spread into the thoracic paravertebral space.

There are different quadratus lumborum blocks (anterior, posterior and lateral blocks) with different mechanisms of action according to injectate spread. However, there is insufficient evidence to recommend one approach and transducer positioning over another for individual patient populations and specific surgical types.

Pericapsular nerve group (PENG) block is relatively a recent regional technique based on blocking the articular branches to the hip joint with a single injection and is used for perioperative analgesia in hip surgery.

The pericapsular nerve group block (PENG) is a regional anesthetic technique described in 2018, developed primarily in total hip arthroplasties (THA) for postoperative analgesia with motor sparing benefits. The block is thought to provide more complete analgesia to the hip by depositing local anesthetic within the myofascial plane of the psoas muscle and superior pubic ramus.

ELIGIBILITY:
Inclusion Criteria:

* Physical status: ASA I-II
* Scheduled for open unilateral hip surgery

Exclusion Criteria:

* Parent's refusal
* Allergy to local anesthetics drugs
* Psychological, mental disorders or metabolic disease
* Patients with bleeding disorder, liver disease or sepsis
* Local infection or pervious surgery at site of anesthetic injection procedures.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
duration of sensory block | within 24 hour postoperative
  It is the time from the end of block performance till the first patient's complain of pain

SECONDARY OUTCOMES:
Pain assessment | immediately postoperative and then at 2, 4, 6, 12 & 24 hours after surgery
  using Modified Objective Pain Scale (MOPS) a scale of 0-10, where 0= No pain and 10= Maximum worst pain.
total amount of post-operative rescue analgesia needed | in the first postoperative 24 hours
  total amount of post-operative rescue analgesia in the form of ibuprofen syrup needed

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Background] Bialik V, Bialik GM, Blazer S, Sujov P, Wiener F, Berant M. Developmental dysplasia of the hip: a new approach to incidence. Pediatrics. 1999 Jan;103(1):93-9. doi: 10.1542/peds.103.1.93. PMID 9917445
- [Background] Gurkan Y, Aksu C, Kus A, Toker K, Solak M. One operator's experience of ultrasound guided lumbar plexus block for paediatric hip surgery. J Clin Monit Comput. 2017 Apr;31(2):331-336. doi: 10.1007/s10877-016-9869-x. Epub 2016 Mar 31. PMID 27033707
- [Background] Kikuchi M, Mihara T, Mizuno Y, Fujimoto H, Arai S, Nomura T, Goto T. Anterior quadratus lumborum block for postoperative recovery after total hip arthroplasty: a study protocol for a single-center, double-blind, randomized controlled trial. Trials. 2020 Feb 5;21(1):142. doi: 10.1186/s13063-020-4090-0. PMID 32024551
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Merella F, Canchi-Murali N, Mossetti V. General principles of regional anaesthesia in children. BJA Educ. 2019 Oct;19(10):342-348. doi: 10.1016/j.bjae.2019.06.003. Epub 2019 Aug 24. No abstract available. PMID 33456856
- [Background] Orozco S, Munoz D, Jaramillo S, Herrera AM. Pediatric use of Pericapsular Nerve Group (PENG) block for hip surgical procedures. J Clin Anesth. 2019 Nov;57:143-144. doi: 10.1016/j.jclinane.2019.04.010. Epub 2019 Apr 22. No abstract available. PMID 31022606